CLINICAL TRIAL: NCT05668039
Title: Enhanced External Counterpulsation (EECP/ECPT) to Treat Long-COVID-19 Fatigue - a Randomized Controlled Trial
Brief Title: Enhanced External Counterpulsation to Treat Long COVID-19 Fatigue
Acronym: EXPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Dafna Yahav, Head, Infectious Diseases Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EECP for long COVID-19
Record Dates: First submitted 2022-12-24; First posted 2022-12-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: long COVID; Enhanced eXternal counterpulsation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Double blind, outcome assossor blind, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking of participants - the sham procedure includes the same location of pneumatic blood-pressure cuffs used for the intervention; and will be perfoemd in the same frequency and duration as the intervention. Participants will be invited for the procedures at separate times to avoid connection between them.
  Masking of investigator and outcome assessor - unblinded nurses and one unblinded physician will be responsible for performing the procedures (either intervention or sham), without involving other team members (other investigators or outcome assessors), who would remain blinded to the treatment arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced external counterpulsation (Experimental): Enhanced external counterpulsation (EECP/ECPT) is a non-invasive technique used to improve cardiac and cerebral perfusion. It aims to achieve 'diastolic augmentation' by increasing arterial blood pressure and retrograde aortic blood flow during diastole. This technique is currently used to treat refractory angina and heart failure, and was demonstrated to be well tolerated without limiting side effect. Practially, blood pressure cuffs are put along the lower limbs and are inflated to 300 mmHg pressure intermittently during one hour session. 15 sessions will be performed over 15 weeks.
  Interventions: Procedure: Enhanced external counterpulsation
- Sham procedure (Sham Comparator): The procedure will be identical to the experimental procedure, excluding the pressure that will reach only 80 mmHg.
  Interventions: Procedure: Enhanced external counterpulsation

INTERVENTIONS:
Procedure: Enhanced external counterpulsation — 15 one-hour sessions during 15 weeks of enhanced external counterpulsation.

SUMMARY:
The goal of this double blind, outcome-assessor blind, randomized controlled trial, is to compare the effectiveness of external encounter counterpulsation (EECP) versus sham procedure in participants with long COVID-19 fatigue.

The main question[s] it aims to answer are:

* Whether EECP improves fatigue score
* Whether EECP improves quality of life, six-minute walk test, and endothelial function Participants will attend 15 sessions (1-hour each) of EECP during 5 weeks Researchers will compare EECP versus sham procedure for the above outcomes.

DETAILED DESCRIPTION:
Participants of this trial will be patients recovering from acute COVID-19, 3-12 months following the acute infection, and suffering from fatigue with a Patient-Reported Outcomes Measurement System (PROMIS)-Fatigue short-form (SF)-7a score of > 50.

Exclusion criteria will include contra-indications for EECP (see protocl). Intervention, comparisn and outcomes are described above. Study plan: participants will be invited using social media, after filling a fatigue score (PROMIS) to test for eligibility. Those with a score of > 50 will be invited for a study visit.

Study visit 1 will include informed consent, followed by physician interview, physical examination, ECG; and will be referred for completion of blood tests including complete blood count (CBC) to rule out significant anemia (Hb< 12 for men or hb <10 for women) and serum beta human chorionic gonadotrophin (bHCG).

Eligible patients will then be randomized into two groups for treatment with EECP vs sham procedure. In study Visit 2 they will answer several questionnaires, perforn EndoPAT test to assess endothelial dysfunction, and six-minute walk test, followed by either:

1. Treatment group- 1 hour EECP session
2. Sham group - 1 hour of a sham EECP session (patients will be hooked to the EECP device but it will be set to the lowest setting, and lowest frequency, therefore unable to create a sufficient rise in diastolic return). This visit will be followed by 3 times weekly 1 hour sessions for 5 weeks (15 sessions) of either EECP or sham procdeure, according to randomization group.

Questionnaire that will be used before and after the intervention will include:

1. Fatigue evaluation using the PROMIS 7a form, attached in appendix (as validated on Myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS)patients)
2. Functional capacity evaluation using the Duke Activity Status Assessment (DASI) (https://www.mdcalc.com/duke-activity-status-index-dasi);
3. Shortness of Breath using the modified Medical Research Council dyspnea scale
4. Quality of life using the SF-36 questionnaire. 6mwt and endothelial dysfunction by EndoPAT will be held following the last treatment.

Study Visit 3 (3 months following starting treatment) will be a final Interview to assess improvement by questionnaires, as well as time to return to activity and time to return to work.

ELIGIBILITY:
Inclusion Criteria:

* Patients recovering from PCR or lateral flow testing proven acute COVID-19
* 3-12 months following the acute infection
* Suffering from fatigue with a PROMIS-SF-7a T-score of > 50

Exclusion Criteria:

* Acute decompensated heart failure
* Recent myocardial infarction within the last 3 months
* Unstable angina pectoris
* Severe hypertension > 180/110 mm Hg
* Coagulopathy with international normalized ratio of prothrombin time > 2.0
* Moderate to severe aortic regurgitation
* Abdominal aortic aneurysm (>5 mm) or dissection
* Arrhythmias that may interfere with triggering of EECP system (uncontrolled atrial fibrillation, flutter and very frequent premature ventricular contractions)
* Heart rate of <35 or >125 beats per minute
* Any surgical intervention within 6 weeks before EECP
* Recent cardiac catheterization (1-2 weeks) or arterial femoral puncture
* Severe peripheral arterial disease
* Severe venous disease (thrombophlebitis, prior or current deep vein thrombosis or pulmonary embolism)
* Severe chronic obstructive pulmonary disease
* Pregnancy or women of childbearing age who do not have a negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue score | 15 weeks
  Change in PROMIS Fatigue 7a T score from baseline. Minimum score is 29, maximum 83, higher levels indicate worse outcome

SECONDARY OUTCOMES:
Change in quality of life score | 15 weeks
  Quality of life improvement per SF-36. Minimum value - 0 and maximum - 100, higher levels indicate worse outcome
Change in six-minute walk test | 15 weeks
  Six-minute walk distance improvement in meters
Cahnge in endothelial function | 15 weeks
  Endothelial dysfunction improvement by EndoPat test

CONTACTS AND LOCATIONS:
Overall Officials: Dana Yelin, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by approaching the PI, with reasonable request

REFERENCES:
- [Background] Michelen M, Manoharan L, Elkheir N, Cheng V, Dagens A, Hastie C, O'Hara M, Suett J, Dahmash D, Bugaeva P, Rigby I, Munblit D, Harriss E, Burls A, Foote C, Scott J, Carson G, Olliaro P, Sigfrid L, Stavropoulou C. Characterising long COVID: a living systematic review. BMJ Glob Health. 2021 Sep;6(9):e005427. doi: 10.1136/bmjgh-2021-005427. PMID 34580069
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Yelin D, Moschopoulos CD, Margalit I, Gkrania-Klotsas E, Landi F, Stahl JP, Yahav D. ESCMID rapid guidelines for assessment and management of long COVID. Clin Microbiol Infect. 2022 Jul;28(7):955-972. doi: 10.1016/j.cmi.2022.02.018. Epub 2022 Feb 17. PMID 35182760
- [Background] Buoite Stella A, Furlanis G, Frezza NA, Valentinotti R, Ajcevic M, Manganotti P. Autonomic dysfunction in post-COVID patients with and witfhout neurological symptoms: a prospective multidomain observational study. J Neurol. 2022 Feb;269(2):587-596. doi: 10.1007/s00415-021-10735-y. Epub 2021 Aug 12. PMID 34386903
- [Background] Fogarty H, Townsend L, Morrin H, Ahmad A, Comerford C, Karampini E, Englert H, Byrne M, Bergin C, O'Sullivan JM, Martin-Loeches I, Nadarajan P, Bannan C, Mallon PW, Curley GF, Preston RJS, Rehill AM, McGonagle D, Ni Cheallaigh C, Baker RI, Renne T, Ward SE, O'Donnell JS; Irish COVID-19 Vasculopathy Study (iCVS) investigators. Persistent endotheliopathy in the pathogenesis of long COVID syndrome. J Thromb Haemost. 2021 Oct;19(10):2546-2553. doi: 10.1111/jth.15490. Epub 2021 Sep 12. PMID 34375505
- [Background] Pretorius E, Vlok M, Venter C, Bezuidenhout JA, Laubscher GJ, Steenkamp J, Kell DB. Persistent clotting protein pathology in Long COVID/Post-Acute Sequelae of COVID-19 (PASC) is accompanied by increased levels of antiplasmin. Cardiovasc Diabetol. 2021 Aug 23;20(1):172. doi: 10.1186/s12933-021-01359-7. PMID 34425843
- [Background] Shechter M, Matetzky S, Feinberg MS, Chouraqui P, Rotstein Z, Hod H. External counterpulsation therapy improves endothelial function in patients with refractory angina pectoris. J Am Coll Cardiol. 2003 Dec 17;42(12):2090-5. doi: 10.1016/j.jacc.2003.05.013. PMID 14680732
- [Background] Bonetti PO, Barsness GW, Keelan PC, Schnell TI, Pumper GM, Kuvin JT, Schnall RP, Holmes DR, Higano ST, Lerman A. Enhanced external counterpulsation improves endothelial function in patients with symptomatic coronary artery disease. J Am Coll Cardiol. 2003 May 21;41(10):1761-8. doi: 10.1016/s0735-1097(03)00329-2. PMID 12767662
- [Background] Varanasi S, Sathyamoorthy M, Chamakura S, Shah SA. Management of Long-COVID Postural Orthostatic Tachycardia Syndrome With Enhanced External Counterpulsation. Cureus. 2021 Sep 30;13(9):e18398. doi: 10.7759/cureus.18398. eCollection 2021 Sep. PMID 34729276
- [Background] Dayrit JK, Verduzco-Gutierrez M, Teal A, Shah SA. Enhanced External Counterpulsation as a Novel Treatment for Post-acute COVID-19 Sequelae. Cureus. 2021 Apr 7;13(4):e14358. doi: 10.7759/cureus.14358. PMID 33987042
- [Background] Yang M, Keller S, Lin JS. Psychometric properties of the PROMIS(R) Fatigue Short Form 7a among adults with myalgic encephalomyelitis/chronic fatigue syndrome. Qual Life Res. 2019 Dec;28(12):3375-3384. doi: 10.1007/s11136-019-02289-4. Epub 2019 Sep 10. PMID 31506915
- [Background] Fan X, Lee KS, Frazier SK, Lennie TA, Moser DK. Psychometric testing of the Duke Activity Status Index in patients with heart failure. Eur J Cardiovasc Nurs. 2015 Jun;14(3):214-21. doi: 10.1177/1474515114523354. Epub 2014 Feb 5. PMID 24504873
- [Background] Rajala K, Lehto JT, Sutinen E, Kautiainen H, Myllarniemi M, Saarto T. mMRC dyspnoea scale indicates impaired quality of life and increased pain in patients with idiopathic pulmonary fibrosis. ERJ Open Res. 2017 Dec 14;3(4):00084-2017. doi: 10.1183/23120541.00084-2017. eCollection 2017 Oct. PMID 29255720
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230